CLINICAL TRIAL: NCT03191448
Title: Evaluation of Healing at Molar Extraction Sites With Ridge Preservation Using Freeze Dried Bone Allograft and a Collagen Wound Dressing
Brief Title: Ridge Preservation Using FDBA and a Collagen Wound Dressing in Molar Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Guy Huynh-Ba, Associate Professor - Clinical, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSC20150708H
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Tooth Extraction

STUDY DESIGN:
Intervention Model Description: This study will document the use of standard care treatment using FDA approved material used in an FDA approved fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ridge preservation in molar sites (Experimental): Patient who will need a single molar site extracted as part of their treatment will be screened and consented for this research study.
  Ridge preservation will be performed in single molar extraction site. The site will be grafted with freezed dried bone allograft (FDBA) and covered with a collagen wound dressing (Collaplug). This is already part of clinical standard care using FDA approved products in an FDA approved fashion. The study aims at documenting the clinical outcome of such accepted procedure more precisely and compare it existing data using other materials.
  Interventions: Procedure: Ridge preservation; Device: FDBA; Device: Collagen wound dressing

INTERVENTIONS:
Procedure: Ridge preservation — Ridge preservation consists of grafting an extraction socket with a bone substitute and /or cover it with a membrane or a dressing. This intervention is aiming at limiting the osseous dimensional changes that would have taken place if the extraction would have been left to heal spontaneously.
  Other Names: Socket preservation; Socket grafting
Device: FDBA — Ridge preservation consists of grafting an extraction socket with a bone substitute and /or cover it with a membrane or a dressing. This intervention is aiming at limiting the osseous dimensional changes that would have taken place if the extraction would have been left to heal spontaneously. In this study a freezed dried bone allograft (FDBA) will be used and the site will be covered with a collagen wound dressing (Collaplug)
Device: Collagen wound dressing — Ridge preservation consists of grafting an extraction socket with a bone substitute and /or cover it with a membrane or a dressing. This intervention is aiming at limiting the osseous dimensional changes that would have taken place if the extraction would have been left to heal spontaneously. In this study a freezed dried bone allograft (FDBA) will be used and the site will be covered with a collagen wound dressing (Collaplug)

SUMMARY:
Currently, it is not known what the dimensional changes might be following a molar site extraction which has been grafted with FDBA and covered with a collagen wound dressing. The purpose of the proposed study is to examine the clinical healing following ridge preservation using freeze dried bone allograft (FDBA) with a collagen wound dressing barrier (CollaPlug®) in a molar extraction site.

I

DETAILED DESCRIPTION:
It is well known that a tooth socket will undergo significant resorption and remodeling following tooth extraction. Pietrokovsky and Massler documented alveolar bone dimension changes subsequent to tooth extraction forty-five years ago. Schropp et al. evaluated tissue changes on models following premolar and molar extractions and concluded that 50% of the ridge width was lost within one year following extraction. Two thirds of this resorption happened during the first 3 months.

In addition to alveolar ridge resorption in a horizontal dimension (decrease in width), changes in the vertical dimension of the ridge have been documented following tooth extraction in a canine model. The healing pattern of the extraction socket observed in the preclinical setting was further confirmed in human investigations). A systematic review concluded that greater loss of ridge width is to be expected following extraction compared to loss of ridge height. Clinical mean reductions of 3.87mm and 1.87mm in ridge width and height, respectively, were reported. Radiographically, the mean reduction amounted 1.21mm and 1.53mm for ridge width and height, respectively. These results were confirmed by another systematic review.

If the extracted tooth is to be replaced, the unfavorable dimensional changes resulting from this healing process may necessitate advanced and technique sensitive guided bone regeneration (GBR) procedures prior to dental implant placement. In order to avoid GBR and limit these dimensional changes, grafting of the extraction socket with or without membrane coverage, also called ridge preservation procedure, have been advocated. In order to perform ridge preservation, typically, a graft material and some sort of a barrier (e.g. non-resorbable and resorbable membranes or collagen wound dressing) are used. A large variety of materials are available on the market for the purpose of ridge preservation. No material gold standard has yet been identified to date, which would ensure the best dimensional stability of the alveolar ridge.

Current materials used as part of standard care in clinical practice include freeze dried bone allograft (FDBA) as a grafting material and a dense polytetrafluroethylene (dPTFE) non-resorbable membrane or a collagen wound dressing (Collaplug®, Zimmer Dental, Carlsbad, CA) to protect the extraction grafted site. It is currently now known how the use of a collagen wound dressing would compare to a non-resorbable membrane (which has been documented) and if any would lead to any substantial clinical advantages.

Therefore, the proposed research project will answer the following question:

What are the dimensional changes of the hard and soft tissues encountered following molar extractions with ridge preservation using FDBA and a collagen wound dressing?

ELIGIBILITY:
Inclusion Criteria:

* One molar tooth that has been identified by dental faculty as requiring a single tooth extraction
* A dental implant is indicated and treatment planned to replace the missing molar tooth
* Have adequate restorative space for a dental implant-retained restoration
* Have at least 10mm of alveolar bone height, without impinging on the maxillary sinus or inferior alveolar canal.

Exclusion Criteria:

* Patients will not be entered who are mentally incompetent, prisoners, or pregnant.
* Pregnant women or women intending to become pregnant during the study period.
* Patients who become pregnant during the study will be withdrawn and standard care will be delivered.
* Clinical and/or radiographic determinations which will preclude inclusion in this study are:

  1. Active localized or systemic infection other than periodontitis.
  2. Untreated periodontal diseases
  3. Inadequate bone dimensions or restorative space dimensions to place a dental implant
  4. Presence of a disease entity, medical condition or therapeutic regimen which decreases probability of soft tissue and bony healing, e.g., poorly controlled diabetes, chemotherapeutic and immunosuppressive agents, or autoimmune diseases.
  5. Positive medical history of endocarditis following oral or dental surgery.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Radiographic bone width changes (in mm) | 3 months
  Following extraction and ridge preservation the alveolar bone around the extraction socket will remodel and some resorption is expected. Alveolar ridge width change (in mm) at the extraction site will be recorded by means of Cone Beam Computed Tomography (CBCT)

SECONDARY OUTCOMES:
Radiographic bone height changes (in mm) | 3 months
  Following extraction and ridge preservation the alveolar bone around the extraction socket will remodel and some resorption is expected. Alveolar ridge height change (in mm) at the extraction site will be recorded by means of Cone Beam Computed Tomography (CBCT)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Araujo MG, Lindhe J. Ridge preservation with the use of Bio-Oss collagen: A 6-month study in the dog. Clin Oral Implants Res. 2009 May;20(5):433-40. doi: 10.1111/j.1600-0501.2009.01705.x. PMID 19522974
- [Background] Barone A, Aldini NN, Fini M, Giardino R, Calvo Guirado JL, Covani U. Xenograft versus extraction alone for ridge preservation after tooth removal: a clinical and histomorphometric study. J Periodontol. 2008 Aug;79(8):1370-7. doi: 10.1902/jop.2008.070628. PMID 18672985
- [Background] Braut V, Bornstein MM, Lauber R, Buser D. Bone dimensions in the posterior mandible: a retrospective radiographic study using cone beam computed tomography. Part 1--analysis of dentate sites. Int J Periodontics Restorative Dent. 2012 Apr;32(2):175-84. PMID 22292147
- [Background] Brownfield LA, Weltman RL. Ridge preservation with or without an osteoinductive allograft: a clinical, radiographic, micro-computed tomography, and histologic study evaluating dimensional changes and new bone formation of the alveolar ridge. J Periodontol. 2012 May;83(5):581-9. doi: 10.1902/jop.2011.110365. Epub 2011 Sep 26. PMID 21942791
- [Background] Darby I, Chen ST, Buser D. Ridge preservation techniques for implant therapy. Int J Oral Maxillofac Implants. 2009;24 Suppl:260-71. PMID 19885449
- [Background] Ferrus J, Cecchinato D, Pjetursson EB, Lang NP, Sanz M, Lindhe J. Factors influencing ridge alterations following immediate implant placement into extraction sockets. Clin Oral Implants Res. 2010 Jan;21(1):22-9. doi: 10.1111/j.1600-0501.2009.01825.x. Epub 2009 Nov 13. PMID 19912273
- [Background] Huynh-Ba G, Pjetursson BE, Sanz M, Cecchinato D, Ferrus J, Lindhe J, Lang NP. Analysis of the socket bone wall dimensions in the upper maxilla in relation to immediate implant placement. Clin Oral Implants Res. 2010 Jan;21(1):37-42. doi: 10.1111/j.1600-0501.2009.01870.x. PMID 20070745
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Background] Nevins M, Camelo M, De Paoli S, Friedland B, Schenk RK, Parma-Benfenati S, Simion M, Tinti C, Wagenberg B. A study of the fate of the buccal wall of extraction sockets of teeth with prominent roots. Int J Periodontics Restorative Dent. 2006 Feb;26(1):19-29. PMID 16515093
- [Background] Oghli AA, Steveling H. Ridge preservation following tooth extraction: a comparison between atraumatic extraction and socket seal surgery. Quintessence Int. 2010 Jul-Aug;41(7):605-9. PMID 20614049
- [Background] Spray JR, Black CG, Morris HF, Ochi S. The influence of bone thickness on facial marginal bone response: stage 1 placement through stage 2 uncovering. Ann Periodontol. 2000 Dec;5(1):119-28. doi: 10.1902/annals.2000.5.1.119. PMID 11885170
- [Background] Tan WL, Wong TL, Wong MC, Lang NP. A systematic review of post-extractional alveolar hard and soft tissue dimensional changes in humans. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:1-21. doi: 10.1111/j.1600-0501.2011.02375.x. PMID 22211303
- [Background] Van der Weijden F, Dell'Acqua F, Slot DE. Alveolar bone dimensional changes of post-extraction sockets in humans: a systematic review. J Clin Periodontol. 2009 Dec;36(12):1048-58. doi: 10.1111/j.1600-051X.2009.01482.x. PMID 19929956
- [Background] Vignoletti F, Matesanz P, Rodrigo D, Figuero E, Martin C, Sanz M. Surgical protocols for ridge preservation after tooth extraction. A systematic review. Clin Oral Implants Res. 2012 Feb;23 Suppl 5:22-38. doi: 10.1111/j.1600-0501.2011.02331.x. PMID 22211304